CLINICAL TRIAL: NCT03931265
Title: Prognostic Evaluations of Ketohexokinase Isoforms in Endometrial Cancer
Brief Title: Ketohexokinase Isoforms in Endometrial Cancer.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 108009-F
Record Dates: First submitted 2019-04-25; First posted 2019-04-30 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ketohexokinase — Check the isoforms of ketohexokinase in the specimen of endometrial cancer

SUMMARY:
Our preliminary analysis with clinical database suggested that, in patients with type I endometrial cancer, high ketohexokinase-expressing group have lower survival probabilities than low ketohexokinase-expressing group. To understand the importance of ketohexokinase expression and isoform switch during the development of type I endometrial cancer, we propose a series of in vitro experiments and clinical examinations in this project.

ELIGIBILITY:
Inclusion Criteria:

* >20 years
* Women with endometrial cancer who are about to be admitted to hospital for gynecological staging.
* Women who have undergone gynecological staging surgery for endometrial cancer in the past.

Exclusion Criteria:

* Women with endometrial cancer who receive preoperative chemotherapy or radiation therapy.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with endometrial cancer who underwent staging surgeries in the Far Eastern Memorial Hospital
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2019-04-11 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The role of ketohexokinase isoforms in the overall survival of endometrial cancer. | 5 years
  Cox proportional hazard regression to evaluate the role of ketohexokinase isoforms in the overall survival of endometrial cancer.

SECONDARY OUTCOMES:
Correlation of ketohexokinase isoforms with the other prognostic risk factors | 5 years
  Correlation of ketohexokinase isoforms with deep myometrial invasion, tumor grade, lymph node metastasis, FIGO stage, tumor size, progression-free survival, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far-Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan